CLINICAL TRIAL: NCT04799236
Title: Treatment of Bolivian Mucosal Leishmaniasis With Miltefosine, Pentavalent Antimony or Liposomal Amphotericin B
Brief Title: Treatment of Mucosal Bolivian Leishmaniasis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion Nacional de Dermatologia (Other)
Collaborators: Hospital Dermatologico de Jorochito (Unknown); Centro Nacional de Enfermedades Tropicales CENETROP (Unknown); ABF Foundation for Medical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABF-BO-2021-100
Record Dates: First submitted 2021-03-09; First posted 2021-03-16 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Mucosal Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Mucocutaneous

STUDY DESIGN:
Intervention Model Description: The primary purpose is to perform a controlled evaluation of the cure rate of miltefosine, LAMB, and Sb for L braziliensis ML in Bolivia.
  A secondary purpose is to determine the tolerance of these regimens.
  Patients will be randomized between:
  Group 1---40 patients. Oral miltefosine. Group 2---40 patients. Intravenous pentavalent antimony (Glucantime) Group 3---40 patients. Intravenous liposomal amphotericin B (Ambisome)
  Because of the disparate routes of administration, the study will not be blinded for the patients or clinical team. However, the ENT doctor who provides data to calculate the primary endpoint, the mucosal severity score, will be blinded.
  After treatment, all patients will be followed for 2, 6, 9, and 12 months after the beginning of therapy. In addition, all attempts will be made to effect follow-up at 24 months.
Who Masked: Investigator
Masking Description: Because of the disparate routes of administration, the study will not be blinded for the patients or clinical team. However, the ENT doctor who provides data to calculate the primary endpoint, the mucosal severity score, will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Oral Miltefosine (Active Comparator): Miltefosine will be administered per os at 150 mg/day [50 mg tid] for 28 days. This is the standard regimen of miltefosine for persons >45 kg.
  Interventions: Drug: Group 1: Miltefosine
- Group 2: Intravenous pentavalent antimony (Active Comparator): IV pentavalent antimony (meglumine antimoniate) will be administrated at 20 mg x kg x d during 20 consecutive days. Antimony will be diluted in 10 times its volume in 5%Dextrose in destilled water and injected IV in 20 minutes
  Interventions: Drug: Group 2: Pentavalent Antimony
- Group 3: Intravenous liposomal amphotericin B (Experimental): LAMB will be administered IV at 3 ampules [150 mg] on each of days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, and 27. Three ampules is the individual dose suggested by Aronson et al [2016] and equals 2.5 mg/kg/dose for a 60 kg person. 15 doses of 3 ampules (total of 2250 mg) equals 37.5 mg/kg for a 60 kg person.
  Interventions: Drug: Group 3: Liposomal amphotericin B

INTERVENTIONS:
Drug: Group 1: Miltefosine — Miltefosine 50 mg pill will be administered po every 8 hours with food, during 28 days
  Arms: Group 1: Oral Miltefosine
Drug: Group 2: Pentavalent Antimony — will be administered by IV infusion diluted in 150 ml of DWD5% over 20 minutes
  Arms: Group 2: Intravenous pentavalent antimony
Drug: Group 3: Liposomal amphotericin B — 3 amps (150 mg) will be administered by IV infusion iver 2 hours every other day for a total of 15 doses.
  Arms: Group 3: Intravenous liposomal amphotericin B

SUMMARY:
The purpose of this protocol is to conduct a randomized comparison of the efficacy and tolerance of miltefosine, LAMB, and pentavalent antimony for the treatment of mucosal leishmaniasis. With such controlled pharmacodynamic data, and additional considerations of administrative convenience (oral >>IV) and cost, we hope that it will be possible for policy makers, treatment professionals, and patients to choose the most appropriate therapy for ML.

ELIGIBILITY:
Inclusion Criteria:

* weight over 45 kg
* Parasitological confirmation of the lesion will be made by visualization of Leishmania, culture of Leishmania, or molecular identification of Leishmania (PCR) from the biopsy or aspirate of the lesion.

Exclusion Criteria:

* Previous treatment for leishmaniasis in the last 12 months
* concomitant diseases by history that would be likely in the PI's opinion to interact, either positively or negatively, with treatment
* values of complete blood count, liver function (aspartate aminotransferase, alkaline phosphatase), renal function (creatinine), pancreatic function (lipase), or uric acid beyond 1.5 x normal range
* EKG with clinically significant abnormalities
* Women of childbearing age not agreeing with the use of secure reproductive contraception for 4 months after initiating miltefosine therapy.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Healing of mucosal lesions | Baseline to 12 month follow up
  The primary purpose is to perform a controlled evaluation of the cure rate of miltefosine, LAMB, and Sb for L braziliensis ML in Bolivia. Using a standarized scale we'll qualify from 0 (absent) to 3 (severe) the following items: erythema, edema/swelling, infiltration, erosion/ulceration, in five different places: nasal and perinasal skin, nasal mucosa, palate and oral mucosa, pharynx and larynx. Additionally, changes in voice quality will be registered. 63 will be the maximun score and means severe and massive compromise.
  clinical cure: >90% loss of presenting severity score clinical improvement: 50%-90% loss of presenting severity score no clinical change: 25% worsening to 49% improvement in presenting severity score clinically worse: >25% worsening of presenting score or relapse after initial improvement

SECONDARY OUTCOMES:
Clinical and laboratory safety of these 3 drugs | Base line to 1 month after the end of therapy
  The secondary purpose is to determine the tolerance of these regimens. Descriptive statistics will be used to present adverse event data. Continuous variables will be presented as number of observations (n), mean, standard deviation (SD), median, minimum and maximum values. Categorical variables will be presented as counts and percentages.
  Adverse effects will be compared between groups by appropriate statistics. During treatment administration clinical symptoms (nausea/vomit/abdominal pain; myalgias/arthralgias; headache/dizziness) and laboratory (AST, alkaline phosphatase, lipase, creatinine, CBC) and EKG (in patients receiving antomony) will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Dermatologico de Jorochito, Santa Cruz de la Sierra, SC, Bolivia